CLINICAL TRIAL: NCT05321446
Title: GoHand(TM) to Enhance Recovery of Arm and Hand Function Post-Stroke
Acronym: GoHand
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Nancy Mayo, James McGill Professor, McGill University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: HBHL Ignite Program 2020
Record Dates: First submitted 2021-10-20; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2021-10

CONDITIONS: Stroke
Keywords: recovery feedback sensors hand function movement
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The intervention is positive auditory feedback provided by the device for good wrist movement during completion of different functional tasks. Two different groups are assessed, one with the device and one without in a sequential pre-post design. The groups are not compared.
Masking Description: No masking required as outcomes are based on technology and performance tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GoHand Feedback Group (Experimental): Both groups will receive a standardized home practice program, the GRASP (Graded Repetitive Arm Supplementary Program). This is a program that has a standard set of arm and hand movements to be practiced 45 minutes per day over a one month period. The person manipulates objects to practice different hand movements. These are everyday objects and each person will be given a set of these to take home and to keep.
  For the Experimental Group, the person will be taught the GRASP program and how to move the wrist and hand optimally to activate the GoHand sensor to hear the sound.
  Interventions: Device: GoHand(TM)
- GoHand Measurement Group (Sham Comparator): For Group 2, the person will be taught GRASP program and how to wear the sensor so it measures movement but does not emit a sound.
  Interventions: Device: GoHand(TM)

INTERVENTIONS:
Device: GoHand(TM) — The GoHand(TM) is a therapeutic wearable that provides positive auditory feedback when the wrist and hand moves optimally during execution of dexterity tests and everyday movements.

SUMMARY:
This is a proof-of-concept study aimed at contributing evidence towards the need, usability and efficacy potential of the GoHandTM sensor in people with reduced hand function post-stroke. A two group, randomized, proof-of-concept, trial. The outcome is change over a one-month period in movement quality as measured by the GoHand sensor. The intervention period is one month. The intervention to be tested is the GoHand sensor, specifically the auditory feedback provided for an optimal wrist and hand movement during everyday tasks. To standardize the practice sessions, all persons will be taught the GRASP (Graded Repetitive Arm Supplementary Program) which has been shown to be of benefit to people recovering from stroke. The intervention group will practice the GRASP program with the sensor in feedback mode and the control group will practice with the sensor without feedback. The total sample size is 12, 6 per group.

The study will be used to create movement metric algorithms and provide preliminary data for extent of change and usability.

DETAILED DESCRIPTION:
Abstract One of the most frustrating and persistent motor sequelae of stroke is poor arm and hand function. There are many therapies for arm function post-stroke. The most effective strategies use repetitive, meaningful movement to promote neuroplasticity to support long lasting improvements in arm function. However, at best, the interventions are only moderately effective in improving impairment related outcomes with little or no carry over into everyday, real-world, activities.

There are two gaps in this area, one is for effective interventions and the second is for methods of measuring outcomes that reflect real-world use of the arm. This study is designed to fill both these gaps with technology. GoHandTM is conceived to be a therapeutic wearable to provide auditory feedback for any voluntary wrist and finger movement. This type of positive auditory feedback is known to stimulate neural connections and, through the process of neural plasticity, imprint the learned movement pattern. The sensor also provides performance feedback that is motivating allowing patients to set and accomplish movement and practice goals and track progress.

The global aim of this project is to develop and validate a sensing and feedback device to the detect disassociated wrist and arm movements and provide auditory feedback for hand movement over a range of starting capacities. The focus is on wrist movement because one of the strongest prognostic indicators for recovery of arm function post-stroke is 20o of active wrist extension and any degree of active finger movement.20 This is a proof-of-concept study aimed at contributing evidence towards the need, usability and efficacy potential of the GoHandTM sensor in people with reduced hand function post-stroke. People with stroke who have arm and hand movement deficits will be invited into a two group, randomized, proof-of-concept, trial. The outcome is change over a one-month period in movement quality as measured by the GoHand sensor. The intervention period is one month. The intervention to be tested is the GoHand sensor, specifically the auditory feedback provided for an optimal wrist and hand movement during everyday tasks. To standardize the practice sessions, all persons will be taught the GRASP (Graded Repetitive Arm Supplementary Program) which has been shown to be of benefit to people recovering from stroke. The intervention group will practice the GRASP program with the sensor in feedback mode and the control group will practice with the sensor without feedback. The total sample size is 12, 6 per group.

The study will be used to create movement metric algorithms and provide preliminary data for extent of change and usability.

ELIGIBILITY:
Inclusion Criteria:

1. Anyone with self-reported difficulties in hand function as indicated by reporting that 2 or more items of the Stroke Impact Scale hand function domain as being somewhat or more difficult to do (as a result of the stroke and not a pre-existing arm problem)
2. Capacity to activate the auditory feedback using the GoHand sensor.

Exclusion Criteria:

1. Stroke more than 2 years ago
2. People who get more than 2/6 items incorrect on the Six-Item Screener.
3. Pain in affected arm that limits mobility and function.
4. Botox in past 3 months for spasticity.
5. People who do not think that they could participate in the prescribed 45 minutes per day of arm and hand activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in hand movement quality metrics from GoHand sensor. | Change over 1 month
  Angular velocity wrist flexion and extension, coefficient of variation, quaterions, while doing standardized dexterity tests (wrist flexion and extension, Box and Block Test, Nine Hole Peg Test) and a set of functional tasks.

SECONDARY OUTCOMES:
Change in Nine Hole Peg Test (NHPT) | Change over 1 month
  The NHPT is administered by asking the participant to take the pegs from a container, one by one, and placing them into the holes on the board, as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container. Participants are scored based on the time taken to complete the test activity, recorded in seconds. Both hands are tested.
Change in Box and Block Test (BBT) | Change over 1 month
  BBT measures unilateral gross manual dexterity. The BBT is composed of a wooden box (53.7 cm x 25.4 cm x 8.5 cm) divided in two compartments by a partition and 150 blocks (2.5 cm). The BBT administration consists of asking the participant to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds. Both hands are tested.
Change in Grip strength | Change over 1 month
  Measured (kg.) for both hands using a hand-held dynamometer (JAMAR).
Change in Stroke Arm Ladder (SF-ARM) | Change over 1 month
  A 20 item index developed using Rasch analysis to measure arm and hand function after stroke. It is classified as a Clinician Reported Outcome (ClinRO) as a clinician rates the quality of movement on an ordinal scale while the participant performs tasks. The SF-ARM measure has been formatted in a manner similar to Computer Adaptive Testing, meaning that the administration of the measure begins at the item representing a middle level of arm and hand function and subsequent items are administered depending on the individuals' responses. In this manner, researchers are able to identify an individuals' exact level of function with the administration of only a fraction of the test items. The result is a shorter, less burdensome and more accurate measure of arm and hand function. The original scoring on a logit scale (-4 to +4) has been transformed to a 0 to 100 scale with 10 points considered clinically meaningful.

OTHER OUTCOMES:
Change in Patient Reported Outcomes | Change over 1 month
  Questionnaires on health aspects of quality of life
Adherence | Over 1 month
  Number and minutes of wear
Change in amount of use | Day 1 and day 30 of home practice period
  Quaterions generated with 12 hours of use on two separate days
Change in Two Minute Walk Test (2MWT) | Change over 1 month
  Distance in meters covered in 2 minutes. Ability to walk is a strong indicator of overall stroke recovery and return to community activities. Poor arm function and walking capacity are linked as engagement of the arm during walking affects muscle activation balance, and trunk rotation.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of the McGill University Health Center, CORE, 5252 de Maisonneuve, Montreal, Quebec, Canada